CLINICAL TRIAL: NCT06513130
Title: Geriatric Assessment at Discharge From the Intensive Care Unit in Patients Aged 75 Years and Older: a Feasibility Study
Acronym: PreGEDI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 9107
Record Dates: First submitted 2024-07-10; First posted 2024-07-22 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Critical Illness; Geriatric Assessment; Older People; Frailty
MeSH Terms: conditions — Critical Illness; Frailty | interventions — Geriatric Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group with geriatric assessment (Experimental): Patients will be assessed by a geriatric physician, in a global (clinical, physical, psyochological and social) approach at the end of the ICU stay or in the 7 days following.
  In addition to the first visit in the group "without geriatric assessment", will be collected:
  * Living conditions (home, proxy, home support)
  * Quality of life (SF-36)
  * Covi test and 4-item Geriatric Depression Scale
  * Katz-ADL and IADL
  * History of fall, mobility assessment
  * Nutritional status (BMI, albuminemia, Mini Nutritionnal Assesment)
  * Cognitive assessment (Mini-mental State Examination)
  The visit at month 6 will be the same in both groups
  Interventions: Other: Geriatric assessment in the 7 days following ICU discharge.
- Group without geriatric assessment (Active Comparator): At the end of the ICU stay or in the 7 days following, will be collect:
  * Medical and surgical history, Charlson comorbidity index,
  * Living place
  * Regular treatment (number and class)
  * ICU trajectory: ICU length of stay, reason for ICU admission, severity scores (SOFA and SAPS 2 score), organ supports requirement and duration
  * Limitation of life-sustaining therapy decision
  At 6 month after ICU discharge, patients will be evaluated during a post-ICU consultation, where will be recorded:
  * Living conditions (home, proxy, home support)
  * Quality of life (SF-36)
  * Covi test and 4-item Geriatric Depression Scale
  * Katz-ADL and IADL
  * History of fall, mobility assessment
  * Nutritional status (BMI, albuminemia, Mini Nutritionnal Assesment)
  * Cognitive assessment (Mini-mental State Examination)
  * Regular treatment (number and class)
  * Hospitalizations between ICU discharge and M6
  * Additional comorbidity
  * Family burden assessment (mini-Zarit)
  Interventions: Other: No geriatric assessment in the 7 days following ICU discharge.

INTERVENTIONS:
Other: Geriatric assessment in the 7 days following ICU discharge. — ICU survivors will be assessed by a geriatric physician, in a global (clinical, physical, psyochological and social) approach at the end of the ICU stay or in the 7 days following ICU discharge.
  Arms: Group with geriatric assessment
Other: No geriatric assessment in the 7 days following ICU discharge. — No geriatric assessment in the 7 days following ICU discharge.
  Arms: Group without geriatric assessment

SUMMARY:
The number of patients aged over 75 continues to grow, and, according to INSEE, will represent almost 10% of the French population in 2021, an increase of 2.4 points since 2000. This demographic change is also observed in the intensive care units, where admitted patients aged over 80 represent now up to 10-20% of critical care admissions, depending on the facility.

The admission of these patients remains controversial, with questions about the benefit to elderly patients, both in terms of in-hospital and distant survival, as well as induced morbidity or subsequent quality of life: functional status is impaired in up to two-thirds of survivors.

The challenge of identifying the patients most able to withstand a stay is a major one. Indeed, a stay in intensive care represents a major stress for the organism, due to the acute condition associated with one or more organ failure(s). Bed rest, immobilization and the use of drugs are responsible for formidable complications in the elderly: muscle-wasting, loss of adaptation to physical effort, loss of autonomy, delirium and agitation, all of which have their own long-term impact.

While many studies have looked at the prognostic factors on admission of these patients, and the selection of the patient with the greatest probability of surviving the intensive care unit (ICU), improving the outcome of patients who survive to the ICU stay remains a little-investigated subject. However, the impact of physical and psychological disturbances induced by these patients' stay in intensive care is major, and their detection and management could be elements of interest in improving the care of this population. However, the feasibility of carrying out such an assessment immediately after an ICU stay has yet to be evaluated. The aim of this study would be to evaluate the feasibility of a geriatric assessment at the end of the ICU stay (or within 7 days of discharge) and at 6 months. This study is a prospective, randomized, single-center, open-label interventional study.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 75 years of age
* Admitted to the intensive care unit, for whatever reason, and having survived their stay, considered as leaving the intensive care unit.
* Subjects affiliated to a health insurance scheme
* Able to understand the aims and risks of the research and to give dated, signed informed consent,
* In the event of confusion on leaving the intensive care unit, a close relative available to give dated, signed informed consent, with the patient's consent collected as soon as his or her condition permits.

Exclusion Criteria:

* Protected subject as defined by law: safeguard of justice, guardianship or curatorship procedures
* Subject moribund, or whose life expectancy as estimated by the clinician in charge is less than 1 month
* Patient not living in Bas-Rhin (visit to M6)

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-01-02 (Estimated); Study Completion 2027-01-02 (Estimated)

PRIMARY OUTCOMES:
Rate of patients for whom a geriatric assessment is carried out between the end of their stay in intensive care and 7 days after discharge. | At 6 Month after ICU discharge

SECONDARY OUTCOMES:
Rate of patients for whom consultation at M6 is carried out. | At 6 Month after ICU discharge
Frailty, assessed using the Clinical Frailty Scale | At 6 Month after ICU discharge
Total hospital length of stay | At 6 Month after ICU discharge
Number of hospitalization | At 6 Month after ICU discharge
Regular treatment modifications | At 6 Month after ICU discharge
  collection of current treatments on admission to intensive care, on discharge from intensive care and hospitalization, and at M6 (prescription)
Modification of place of living | At 6 Month after ICU discharge
  location (single-family dwelling, retirement home, etc.)
Evolution of the quality of life assessed by the SF-36 questionnary | At 6 Month after ICU discharge
  For the interventional arm
Evolution of the psychological behaviours through the mini Geriatric depression score evolution and the Covi test evolution for the anxiety component. | At 6 Month after ICU discharge
  For the interventional arm
Evolution of the psychological behaviours through the Covi test evolution for the anxiety component. | At 6 Month after ICU discharge
  For the interventional arm
Evolution of the Katz-ADL score between initial assessment and month 6 | At 6 Month after ICU discharge
  For the interventional arm For the control arm,
Evolution of the IADL score between initial assessment and month 6 | At 6 Month after ICU discharge
  For the interventional arm For the control arm,
Evolution of the locomotor abilities | At 6 Month after ICU discharge
Evolution of cognition evaluation: mini Mental State Examination | At 6 Month after ICU discharge
At M6: main organ function assessment | At 6 Month after ICU discharge

CONTACTS AND LOCATIONS:
Overall Officials: Julien DEMISELLE, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de Médecine Intensive - Réanimation / CHU Strasbourg - France, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No